CLINICAL TRIAL: NCT05786911
Title: Evaluation of Postpartum Fatigue and Pain, After Childbirth Under Epidural Analgesia, According to the Nutritional Status of the Parturient: A Monocentric Observational Prospective Study
Brief Title: Postpartum Fatigue and Pain Versus Nutritional Status, With Epidural Analgesia
Status: Completed | Type: Observational
Sponsor: CHU de Charleroi (Other)
Collaborators: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Maïté Beugnies, Principal Investigator Doctor Beugnies Maïté, CHU de Charleroi
Other Study IDs: P2022/271,B406202200014
Record Dates: First submitted 2023-03-05; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Vaginal Delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- vaginal delivery under epidural: 60 patients, having had a vaginal delivery under an epidural, will be recruited at the maternity ward
  Interventions: Other: nutritional score

INTERVENTIONS:
Other: nutritional score — correlation between a food habit and nutritional status score of the parturient and a postpartum fatigue (FSS) and pain (ENA) score

SUMMARY:
The objective of this preliminary observational study is to evaluate, in the patient, a correlation between a food habit and nutritional status score of the parturient and a postpartum fatigue (FSS) and pain (ENA) score on day 1, 3 and 7.

DETAILED DESCRIPTION:
Several studies, focusing on nutrition during pregnancy, show that a healthy diet during pregnancy promotes fetal growth and development and has been associated with lower risks of complications, while unhealthy diets, undernutrition and overeating have been associated with adverse effects. Indeed, the FIGO initiative developed in 2015 a short nutritional questionnaire on adolescent nutrition, preconception and mothers. The FIGO Nutrition Checklist is an acceptable, potentially feasible, and validated clinical practice tool that can identify regular consumption of unhealthy diets or other nutrition and weight-related issues.

Studies have shown that exhaustion, fatigue and pain are commonly experienced by the mother during the postpartum period and can impact daily functioning, mental health and parenting practices.

Currently, the link between nutritional status, eating habits and postpartum pain and fatigue has not yet been clearly studied. Recognizing patients at risk of pain and fatigue, due to their nutritional status, could make it possible to adapt and anticipate their treatment, in particular analgesics, and to consider multidisciplinary management.

The objective of this preliminary observational study is to evaluate, in the patient, a correlation between a score of eating habits and nutritional status of the parturient and a score of fatigue and postpartum pain at D 1, 3. and 7.

After obtaining written consent, 60 patients, having given birth vaginally under an epidural, will be recruited at the maternity ward. The exclusion criteria will be the patient's refusal, the absence of communication in French, the impossibility of giving free and informed consent, surgery under anesthesia during hospitalization.

Questionnaires adapted to assess the nutritional score and the PNNS-GS 2 eating habits of the patients will be completed by the doctor, at the maternity ward on D 1 postpartum. To do this, a typical 24-hour food day will be harvested and then extrapolated to a week. Age, lifestyle, sports habits, vitamin intake before and during pregnancy, weight before and during pregnancy, height, BMI, ASA status, history, duration of labour, complications during pregnancy, complications during childbirth, tears of the perineum, biology data and analgesic treatments will be collected in the medical file. A fatigue and pain score, FSS score and ENA score, respectively at rest and in motion, will be completed by the doctor on D1, D3 and D7 postpartum, either at the maternity ward or by telephone contact. The differences between the scores of days 1, 3 and 7 will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* vaginal delivery under epidural

Exclusion Criteria:

* patient's refusal
* lack of communication in French
* inability to give free and informed consent
* surgery under anesthesia during hospitalization

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — eligibility is based on female gender: inclusion criteria vaginal delivery under epidural
Study Population: Female population of age to carry a pregnancy to term, with an uncomplicated vaginal delivery under epidural analgesia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
PNNSGS2 | day 1
  nutrition score
ENA: analog digital scale | day 1
  Analog pain scale: 0 no pain and 10 worst pain
ENA: analog digital scale | day 3
  Analog pain scale: 0 no pain and 10 worst pain
ENA: analog digital scale | day 7
  Analog pain scale: 0 no pain and 10 worst pain
FSS: Fatigue Severity Scale | day 1
  fatigue score: 0 not tired and 10 very tired
FSS: Fatigue Severity Scale | day 3
  fatigue score: 0 not tired and 10 very tired
FSS: Fatigue Severity Scale | day 7
  fatigue score: 0 not tired and 10 very tired

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PD Dony, PhD, Study Director — CHU de Charleroi
Locations (1):
- CHU de Charleroi, Charleroi, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No
We do not yet know if the IPD sharing plan will be implemented

REFERENCES:
- [Background] Valko PO, Bassetti CL, Bloch KE, Held U, Baumann CR. Validation of the fatigue severity scale in a Swiss cohort. Sleep. 2008 Nov;31(11):1601-7. doi: 10.1093/sleep/31.11.1601. PMID 19014080
- [Background] Chaltiel D, Adjibade M, Deschamps V, Touvier M, Hercberg S, Julia C, Kesse-Guyot E. Programme National Nutrition Sante - guidelines score 2 (PNNS-GS2): development and validation of a diet quality score reflecting the 2017 French dietary guidelines. Br J Nutr. 2021 Jan 14;125(1):118-120. doi: 10.1017/S0007114520004134. No abstract available. PMID 33319724
- [Background] Tsoi KY, Chan RSM, Li LS, McAuliffe FM, Hanson MA, Tam WH, Ma RCW. Evaluation of dietary pattern in early pregnancy using the FIGO Nutrition Checklist compared to a food frequency questionnaire. Int J Gynaecol Obstet. 2020 Sep;151 Suppl 1(Suppl 1):37-44. doi: 10.1002/ijgo.13324. PMID 32894588
- [Background] McAuliffe FM, Killeen SL, Jacob CM, Hanson MA, Hadar E, McIntyre HD, Kapur A, Kihara AB, Ma RC, Divakar H, Hod M. Management of prepregnancy, pregnancy, and postpartum obesity from the FIGO Pregnancy and Non-Communicable Diseases Committee: A FIGO (International Federation of Gynecology and Obstetrics) guideline. Int J Gynaecol Obstet. 2020 Sep;151 Suppl 1(Suppl 1):16-36. doi: 10.1002/ijgo.13334. No abstract available. PMID 32894590
- See also: Factors associated with maternal postpartum fatigue: an observationalstudy — https://bmjopen.bmj.com/content/9/7/e025927
- See also: Overview of the postpartum period: Normal physiology and routine maternal care — https://www.medilib.ir/uptodate/show/6711
- See also: Overview of the postpartum period: Disorders and complications — https://www.medilib.ir/uptodate/show/127985
- See also: Nutrition in pregnancy: Assessment and counseling — https://www.medilib.ir/uptodate/show/130920